CLINICAL TRIAL: NCT00248040
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group Pilot Study to Assess Efficacy, Safety and Pharmacokinetics of 2 Schedules of Reparixin in the Prevention of Delayed Graft Function After Kidney Transplant in High Risk Patients
Brief Title: Reparixin in Prevention of Delayed Graft Function After Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REP0204
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2020-09

CONDITIONS: Ischemia-Reperfusion Injury; Kidney Diseases
Keywords: Kidney transplantation; Reperfusion Injury; Survival
MeSH Terms: conditions — Reperfusion Injury; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- reparixin group - continuous infusion (Experimental): Continuous iv infusion into a (high flow) central vein (or through an arterio-venous fistula) by an infusion pump.
  A dose of 2.772 mg/kg/h was administered for12 hours.
  Interventions: Drug: Reparixin continuous infusion
- reparixin group - intermittent infusion (Experimental): Intermittent iv infusion into a (high flow) central vein (or through an arterio-venous fistula) by an infusion pump.
  A dose of 2.244 mg/kg was administered over a 30-minute period, followed by a 1.5-hour interval. Twelve doses were administered over a total period of 22.5 hours.
  Interventions: Drug: reparixin intermittent infusion
- placebo infusion (Placebo Comparator): Continuous/intermittent iv infusion of a volume/schedule matched saline into a (high flow) central vein (or through an arterio-venous fistula) by an infusion pump.
  Interventions: Other: placebo infusion

INTERVENTIONS:
Drug: Reparixin continuous infusion — The Investigational Product was administered as an intravenous infusion into a (high flow) central vein or through an arterio-venous fistula, by an infusion pump adequate to provide reliable infusion rates, as per treatment schedule. Total infusion volume did not exceed 500 mL/24 hours. A dose of 2.772 mg/kg body weight/hour was to be administered for 12 hours. Placebo was volume/schedule matched saline.
  Other Names: REP
  Arms: reparixin group - continuous infusion
Drug: reparixin intermittent infusion — A dose of 2.244 mg/kg body weight was to be administered over a 30-minute period, followed by a 1.5-hour interval. Twelve doses were to be administered over a total period of 22.5 hours. Placebo was volume/schedule matched saline.
  Other Names: REP
  Arms: reparixin group - intermittent infusion
Other: placebo infusion — placebo was volume/schedule matched saline
  Arms: placebo infusion

SUMMARY:
The chemokine CXCL8 plays a key role in the recruitment and activation of polymorphonuclear neutrophils in post-ischemia reperfusion injury after solid organ transplantation. Reparixin is a novel, specific inhibitor of CXCL8. This study is configured to explore the safety and efficacy of reparixin in preventing the delayed graft function (DGF) after kidney transplantation.

DETAILED DESCRIPTION:
Delayed graft function (DGF) is the most common allograft complication in the immediate kidney post-transplant period, affecting 25-35% of all patients who receive a cadaver graft, but rates up to 50% have been reported, especially in recipients of kidneys from marginal donors. It is an important clinical complication as it requires dialysis, prolongs hospitalisation, raises the cost of transplantation, and makes more difficult the management of immunosuppressive therapy. Although the effects of DGF on long-term graft function are still debated, there is overall increasing evidence that DGF reduces long-term graft survival. Moreover, given the well documented impact of acute rejection on long-term graft survival, it is conceivable that DGF and acute rejection synergize in negatively influencing long-term graft survival. Kidney reperfusion, after long cold ischemia period, is associated with an inflammatory reaction characterized by massive polymorphonuclear leukocyte (PMN) infiltration both at the glomerular and tubular levels. The importance of CXCL8 in recruiting PMN in kidney tissue during the ischemic time and after reperfusion has been clearly documented.

The efficacy of reparixin in preventing PMN infiltration and tissue damage in rat models of kidney transplantation and lung transplantation, as well as the safety shown in human phase 1 studies, provide the rationale for a clinical study aimed at evaluating the effect of reparixin in preventing DGF after kidney transplantation

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients accepted and listed for renal transplantation due to end stage renal disease (ESRD)
* Planned isolated single kidney transplant from a non-living donor with brain death
* Recipients of a kidney maintained in cold storage
* Recipients at risk of developing DGF
* Planned induction with steroids + mycophenolate mofetil (MMF) or mycophenolic acid + biological induction
* Patient willing and able to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations
* Patient given written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care

Exclusion Criteria:

* Recipients of an intended multiple organ transplant
* Recipients of a kidney from a living donor
* Recipients of a kidney from a non-heart beating donor
* Recipients of double kidney transplant
* Re-transplant >2
* Recipients of a kidney maintained by pulsatile machine perfusion
* Concurrent sepsis
* Recipients with hepatic dysfunction at the time of transplant
* Clinical contraindications to central line access, or arteriovenous fistula, if any, not suitable for infusion of investigational product
* Hypersensitivity to non steroidal anti-inflammatory drugs (NSAIDs)
* Patients simultaneously participating in any other clinical trials involving an investigational drug not yet authorized for use in kidney transplant
* Pregnant or breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII
Locations (9):
- United States (2):
  - Transplant Center, University of Minnesota Medical School, Minneapolis, Minnesota
  - Division of Transplantation, Drexel University College of Medicine, Philadelphia, Pennsylvania
- France (2):
  - Service de Nephrologie et Transplantation, Hopital Lapeyronie, Centre Hospitalier Universitaire Montpellier, Montpellier
  - Service de Transplantation et Soins Intensifs Nephrologiques, Hopital Necker, Paris
- Italy (3):
  - Divisione di Nefrologia e Dialisi, Ospedali Riuniti di Bergamo, Bergamo
  - Divisione di Nefrologia e Dialisi, Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Università degli Studi di Padova, Clinica Chirurgica III, Padua
- Spain (2):
  - Renal Transplant Unit, Hopital Clinic i Provincial de Barcelona, Barcelona
  - Division of Nephrology, Institut Catala de la Salut, Ciutat Sanitaria i Universitaria de Bellvitge, Barcelona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 74 pt. (25 & 23 in reparixin continuous and intermittent infusion, and 26 in the pooled placebo) received the drug and were included in the safety population; 73 pt. (24, 23, 26) received both the study drug and the transplant and were included in the ITT. 1 started study drug but did not receive a kidney transplant, so was excluded from the ITT.
Pre-assignment Details: Six patients (2 in the reparixin continuous infusion group; 3 in the reparixin intermittent infusion group; 1 in the placebo intermittent infusion group) did not receive Investigational Product(s) or kidney transplants and hence they were excluded from both the Safety and ITT populations.
Groups:
- Reparixin Continuous Infusion: Continuous iv infusion into a (high flow) central vein (or through an arterio-venous fistula) by an infusion pump.
  A dose of 2.772 mg/kg/h was administered for12 hours.
- Reparixin Intermittent Infusion: Intermittent iv infusion into a (high flow) central vein (or through an arterio-venous fistula) by an infusion pump.
  A dose of 2.244 mg/kg was administered over a 30-minute period, followed by a 1.5-hour interval. Twelve doses were administered over a total period of 22.5 hours.
- Placebo Continuous/Intermittent Infusion: Continuous/intermittent iv infusion of a volume/schedule matched saline into a (high flow) central vein (or through an arterio-venous fistula) by an infusion pump.
Period: Overall Study
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Started | 25 | 23 | 26
Completed | 22 | 22 | 22
Not Completed | 3 | 1 | 4
Not completed — transplantectomy | 2 | 1 | 3
Not completed — transplant cancelled post treat start | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion | Total
Number analyzed (Participants) | 25 | 23 | 26 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 23 | 26 | 74
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (7.4) | 55.9 (6.3) | 51.4 (11.3) | 53.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 19 | 50
  Male | 7 | 10 | 7 | 24
Region of Enrollment [Number; unit: participants]
  France | 10 | 9 | 10 | 29
  United States | 2 | 2 | 4 | 8
  Spain | 7 | 5 | 4 | 16
  Italy | 6 | 7 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Creatinine Clearance (CrCl) in the Immediate Post-transplant Period
Description: CrCl was determined by two 60 minute urine collections, during the time intervals 1-3 and 10-12 hours of allograft reperfusion. Blood was withdrawn at the midpoint of each urine collection. CrCl at each timepoint was calculated according to the formula:
  creatinine clearance (mL/minutes) = urine creatinine (mmol/L) x urine volume (mL) / serum creatinine (mmol/L) x time of collection (minutes) An average was to be calculated from the two 60 minute values in each interval.
Time Frame: 1-3 and 10-12 hours post allograft reperfusion
Population: ITT population. The ITT population consisted of all randomized patients who received any Investigational Product(s) and a kidney transplant.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
mL/min
  1-3 hours post-transplant: number analyzed (Participants) | 21 | 20 | 23
  1-3 hours post-transplant | 5.11 (8.56) | 7.44 (12.81) | 6.30 (6.26)
  10-12 hours post-transplant: number analyzed (Participants) | 21 | 21 | 20
  10-12 hours post-transplant | 9.66 (10.52) | 14.45 (17.39) | 10.75 (10.93)
Statistical Analysis 1: Comparison: Reparixin Continuous Infusion vs Placebo Continuous/Intermittent Infusion; This analysis refers to the 1-3 hours time point; Test type: Superiority — The model included fixed effect terms for center, time point, and treatment. Time point was specified as a repeated measurement; p = 0.9076, Other; Difference between means = -0.275, 95% CI 2-sided [-5.00 to 4.45]
Statistical Analysis 2: Comparison: Reparixin Intermittent Infusion vs Placebo Continuous/Intermittent Infusion; This analysis refers to the 1-3 hours timepoint; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3084, Other; Difference between means = 2.444, 95% CI 2-sided [-2.32 to 7.21]
Statistical Analysis 3: Comparison: Reparixin Continuous Infusion vs Reparixin Intermittent Infusion; Test type: Other; p = 0.2565, Other; Difference between means = -2.719, 95% CI 2-sided [-7.47 to 2.03]
Statistical Analysis 4: Comparison: Reparixin Continuous Infusion vs Placebo Continuous/Intermittent Infusion; This analysis refers to the 10-12 hours time point; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9855, Other; Difference between means = -0.063, 95% CI 2-sided [-6.91 to 6.79]
Statistical Analysis 5: Comparison: Reparixin Intermittent Infusion vs Placebo Continuous/Intermittent Infusion; This analysis refers to the 10-12 hours timepoint; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1934, Other; Difference between means = 4.519, 95% CI 2-sided [-2.36 to 11.39]
Statistical Analysis 6: Comparison: Reparixin Continuous Infusion vs Reparixin Intermittent Infusion; This analysis refers to the 10-12 hours time point; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1797, Other; Difference between means = -4.582, 95% CI 2-sided [-11.3 to 2.17]

2. Secondary Outcome: Renal Function Tests - Serum Creatinine
Description: Serum creatinine (SrCr) was measured daily from Day 1 up to 7 days post-transplant or up to hospital discharge, whichever occurred earlier; in patients undergoing dialysis, SrCr values were measured immediately before dialysis.
Time Frame: daily up to day 7 post-transplant or hospital discharge
Population: The ITT population consisted of all randomized patients who received any Investigational Product(s) and a kidney transplant.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Infusion
Number analyzed (Participants) | 24 | 23 | 26
mmol/L
  Day 1: number analyzed (Participants) | 24 | 22 | 23
  Day 1 | 0.686 (0.178) | 0.643 (0.219) | 0.651 (0.202)
  Day 2: number analyzed (Participants) | 24 | 23 | 25
  Day 2 | 0.683 (0.244) | 0.576 (0.254) | 0.658 (0.278)
  0.Day 3: number analyzed (Participants) | 24 | 23 | 25
  0.Day 3 | 0.632 (0.311) | 0.500 (0.270) | 0.613 (0.317)
  Day 4: number analyzed (Participants) | 24 | 23 | 25
  Day 4 | 0.589 (0.330) | 0.427 (0.260) | 0.601 (0.360)
  Day 5: number analyzed (Participants) | 24 | 23 | 25
  Day 5 | 0.509 (0.281) | 0.383 (0.253) | 0.567 (0.367)
  Day 6: number analyzed (Participants) | 24 | 23 | 25
  Day 6 | 0.510 (0.334) | 0.333 (0.206) | 0.570 (0.407)
  Day 7: number analyzed (Participants) | 24 | 23 | 25
  Day 7 | 0.474 (0.351) | 0.318 (0.212) | 0.542 (0.411)

3. Secondary Outcome: Renal Function Tests - Calculated Glomerular Filtration Rate
Description: Calculated glomerular filtration rate (GFR) was measured daily from Day 1 up to 7 days post-transplant or up to hospital discharge, whichever occurred earlier; in patients undergoing dialysis, SrCr values were measured immediately before dialysis
Time Frame: from Day 1 up to 7 days post-transplant or up to hospital discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
mL/min
  Day 1: number analyzed (Participants) | 24 | 22 | 23
  Day 1 | 6.04 (2.99) | 8.03 (6.46) | 7.03 (3.48)
  Day 2: number analyzed (Participants) | 24 | 23 | 25
  Day 2 | 6.95 (5.00) | 10.68 (8.61) | 8.74 (8.06)
  Day 3: number analyzed (Participants) | 24 | 23 | 25
  Day 3 | 10.99 (12.26) | 14.86 (11.67) | 13.15 (15.22)
  Day 4: number analyzed (Participants) | 24 | 23 | 25
  Day 4 | 13.90 (15.15) | 19.64 (15.28) | 15.79 (18.57)
  Day 5: number analyzed (Participants) | 24 | 23 | 25
  Day 5 | 17.97 (22.53) | 23.91 (19.02) | 18.61 (22.03)
  Day 6: number analyzed (Participants) | 24 | 23 | 25
  Day 6 | 20.46 (24.24) | 26.64 (19.81) | 20.75 (24.01)
  Day 7: number analyzed (Participants) | 24 | 23 | 25
  Day 7 | 22.42 (22.35) | 28.06 (20.10) | 22.70 (24.45)

4. Secondary Outcome: Renal Function Tests - Urine Output
Description: Urine output, measured in the interval from transplant to 8:00 of Day 1, and then daily from Day 2 up to 7 days post-transplant or up to hospital discharge, whichever occurred earlier
Time Frame: from Day 1 up to 7 days post-transplant or up to hospital discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
mL
  Day 1: number analyzed (Participants) | 24 | 22 | 25
  Day 1 | 1615.9 (2082.7) | 1749.9 (2109.9) | 1925.3 (2214.1)
  Day 2: number analyzed (Participants) | 24 | 22 | 25
  Day 2 | 2242.7 (2236.8) | 2620.2 (2444.1) | 2844.5 (2861.2)
  Day 3: number analyzed (Participants) | 24 | 22 | 25
  Day 3 | 2321.1 (2087.8) | 2979.6 (2000.1) | 2904.0 (2468.3)
  Day 4: number analyzed (Participants) | 24 | 23 | 25
  Day 4 | 2409.8 (2043.2) | 2583.3 (1698.6) | 2939.4 (2585.0)
  Day 5: number analyzed (Participants) | 24 | 23 | 25
  Day 5 | 1958.2 (1609.2) | 2474.8 (1575.4) | 2035.4 (1816.7)
  Day 6: number analyzed (Participants) | 24 | 23 | 25
  Day 6 | 1795.8 (1206.2) | 2239.3 (1228.1) | 1994.8 (1688.5)
  Day 7: number analyzed (Participants) | 24 | 23 | 25
  Day 7 | 2072.3 (1240.9) | 2226.1 (1093.2) | 1805.1 (1390.9)

5. Secondary Outcome: Number of Patients Requiring Dialysis Within 7 Days Post-transplant
Description: The number of patients who required dialysis within 7 days post-transplant was evaluated.
Time Frame: up to day 7 post-transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Infusion
Number analyzed (Participants) | 24 | 23 | 26
Participants
  Yes | 7 | 7 | 6
  No | 15 | 15 | 18
  Unknown | 2 | 1 | 2

6. Secondary Outcome: Number of Days on Dialysis Before Resuming Kidney Function
Description: the number of days on dialysis before resuming kidney function was evaluated.
Time Frame: up to Day 7 post-transplant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
days | 2.5 (0.7) | 1.0 (0.0) | 2.0 (0.0)

7. Secondary Outcome: Number of Patients With Immediate, Slow and Delayed Graft Function
Description: The number of patients who required dialysis within 7 days post-transplant was evaluated.
  Immediate graft function: SrCr ≤3 mg/dL on post operative day 5) Slow graft function: SrCr >3 mg/dL dL on post operative day 5, no need of dialysis) Delayed graft function: Dialysis needed in the first week)
Time Frame: day 5 post-transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
Participants
  Immediate graft function | 6 | 10 | 7
  Slow graft function | 8 | 5 | 11
  Delayed graft function | 8 | 8 | 6
  Unknown | 2 | 0 | 2

8. Secondary Outcome: Duration of Hospital Stay
Description: The mean duration of hospital stay was evaluated.
Time Frame: first 30 days post-transplant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
days | 14.6 (8.4) | 16.1 (7.6) | 13.3 (7.9)

9. Secondary Outcome: Mortality
Description: Mortality in the first 30 days post-transplant was evaluated.
Time Frame: first 30 days post-transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
Participants
  No | 24 | 23 | 25
  Yes | 0 | 0 | 1

10. Secondary Outcome: Serum Creatinine at Month 1, Month 6 and Month 12
Description: Serum creatinine (SrCr) was measured at Month 1, Month 6 and Month 12.
Time Frame: at Month 1, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmo/L
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
mmo/L
  Month 1: number analyzed (Participants) | 22 | 22 | 22
  Month 1 | 0.252 (0.2250) | 0.169 (0.0777) | 0.186 (0.0890)
  Month 6: number analyzed (Participants) | 19 | 22 | 21
  Month 6 | 0.145 (0.0658) | 0.139 (0.0417) | 0.179 (0.1227)
  Month 12: number analyzed (Participants) | 19 | 21 | 21
  Month 12 | 0.150 (0.0879) | 0.150 (0.0618) | 0.227 (0.2578)

11. Secondary Outcome: Calculated Serum Creatinine Clearance at Month 1, Month 6 and Month 12
Description: Creatinine clearance (CrCl) is the volume of blood plasma cleared of creatinine per unit time. It is a rapid and cost-effective method for the measurement of renal function.
Time Frame: at Month 1, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
mL/min
  Month 1: number analyzed (Participants) | 22 | 22 | 21
  Month 1 | 42.86 (22.56) | 44.75 (16.20) | 41.21 (14.23)
  Month 6: number analyzed (Participants) | 19 | 21 | 20
  Month 6 | 52.43 (18.18) | 51.14 (12.54) | 46.93 (16.65)
  Month 12: number analyzed (Participants) | 19 | 21 | 21
  Month 12 | 53.48 (20.39) | 51.10 (15.07) | 41.74 (19.03)

12. Secondary Outcome: Acute Rejection Episodes at Month 6 and Between Month 6 and Month 12
Description: Acute rejection defined as an increase in serum creatinine level after exclusion of other causes of graft dysfunction, accompanied by a sudden decline in glomerular filtration rate and renal function and well-established diagnostic features on kidney allograft biopsy which can be either antibody-mediated and/or T cell-mediated and can occur at any time after transplant.
Time Frame: at Month 6 and between Month 6 and Month 12
Population: as for outcome 2
Measure: Number; unit: episodes
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
episodes
  Month 6 | 2 | 6 | 2
  Between Month 6 and Month 12 | 0 | 0 | 4

13. Secondary Outcome: Patient Survival Rate
Description: Numbers of patients alive, dead, and lost to follow up are reported.
Time Frame: at Month 1, Month 6 and Month 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
Participants
  Month 1 - Alive | 22 | 22 | 22
  Month 1 - Dead | 0 | 0 | 1
  Month 1 - Lost to follow up | 2 | 1 | 3
  Month 6 - Alive: number analyzed (Participants) | 22 | 22 | 22
  Month 6 - Alive | 20 | 22 | 21
  Month 6 - Dead: number analyzed (Participants) | 22 | 22 | 22
  Month 6 - Dead | 0 | 0 | 0
  Month 6 - Lost to follow up: number analyzed (Participants) | 22 | 22 | 22
  Month 6 - Lost to follow up | 2 | 0 | 1
  Month 12 - Alive: number analyzed (Participants) | 20 | 22 | 21
  Month 12 - Alive | 19 | 21 | 21
  Month 12 - Dead: number analyzed (Participants) | 20 | 22 | 21
  Month 12 - Dead | 0 | 1 | 0
  Month 12 - Lost to follow up: number analyzed (Participants) | 20 | 22 | 21
  Month 12 - Lost to follow up | 1 | 0 | 0

14. Secondary Outcome: Graft Survival Rate
Description: Graft failure was defined as the failure of graft function for any reason, ultimately requiring renal replacement therapy and/or retransplantation (United States Renal Data System [USRDS] 2017.
Time Frame: at Month 1, Month 6 and Month 12
Population: as for outcome 2
Measure: Number; unit: number of grafts
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
Number analyzed (Participants) | 24 | 23 | 26
number of grafts
  Month 1 - Graft functioning: number analyzed (Participants) | 24 | 23 | 25
  Month 1 - Graft functioning | 21 | 22 | 22
  Month 1 - Graft failed: number analyzed (Participants) | 24 | 23 | 25
  Month 1 - Graft failed | 3 | 1 | 3
  Month 6 - Graft functioning: number analyzed (Participants) | 19 | 22 | 21
  Month 6 - Graft functioning | 19 | 22 | 20
  Month 6 - Graft failed: number analyzed (Participants) | 19 | 22 | 21
  Month 6 - Graft failed | 0 | 0 | 1
  Month 12 - Graft functioning: number analyzed (Participants) | 19 | 21 | 20
  Month 12 - Graft functioning | 18 | 20 | 20
  Month 12 - Graft failed: number analyzed (Participants) | 19 | 21 | 20
  Month 12 - Graft failed | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: All AEs were reported up to 10 days or hospital discharge. Thereafter, only untoward events that the Investigator assessed as at least possibly related to the study drug were recorded
Arm/Group | Reparixin Continuous Infusion | Reparixin Intermittent Infusion | Placebo Continuous/Intermittent Infusion
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 1/26
Serious Adverse Events (participants affected / at risk) | 12/25 | 5/23 | 9/26
Other Adverse Events (participants affected / at risk) | 24/25 | 23/23 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin Continuous Infusion (N=25) | Reparixin Intermittent Infusion (N=23) | Placebo Continuous/Intermittent Infusion (N=26)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PERIRENAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
URINARY ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL VEIN THROMBOSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
URETERIC FISTULA (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
RENAL ARTERY THROMBOSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
COMPLICATIONS OF TRANSPLANTED KIDNEY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URETERAL NECROSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
RETROPERITONEAL HAEMORRHAGE (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin Continuous Infusion (N=25) | Reparixin Intermittent Infusion (N=23) | Placebo Continuous/Intermittent Infusion (N=26)
ANAEMIA (Blood and lymphatic system disorders) | 6 (6) | 10 (10) | 12 (12)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
BLEPHARITIS (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 8 (8) | 5 (5) | 6 (6)
VOMITING (Gastrointestinal disorders) | 5 (5) | 1 (1) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 1 (1) | 4 (4)
OEDEMA (General disorders) | 2 (2) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 2 (2) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 2 (2) | 0 (0)
HAEMORRHAGIC CYST (General disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 0 (0) | 2 (2) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4) | 5 (5) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COMPLICATIONS OF TRANSPLANTED KIDNEY (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FEMORAL NERVE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PERINEPHRIC COLLECTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PERIRENAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RENAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
URINARY ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BLOOD PHOSPHORUS INCREASED (Investigations) | 1 (1) | 0 (0) | 2 (2)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD AMYLASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 4 (4)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (4) | 6 (6) | 3 (3)
ACIDOSIS (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 5 (5)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 4 (4)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 3 (3) | 2 (2) | 3 (3)
ANXIETY (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 5 (5) | 7 (7) | 7 (7)
BLADDER SPASM (Renal and urinary disorders) | 4 (4) | 2 (2) | 1 (1)
ANURIA (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
RENAL VEIN THROMBOSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
URETERIC FISTULA (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
RENAL INFARCT (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
BLADDER PAIN (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OLIGURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL TUBULAR DISORDER (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URETERAL NECROSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY BLADDER ATROPHY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URINOMA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
METRORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
SCROTAL OEDEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
COMPLICATIONS OF TRANSPLANTED KIDNEY (Renal and urinary disorders) | 3 (3) | 0 (0) | 4 (4)
RENAL ARTERY THROMBOSIS (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
BRADYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 6 (6) | 5 (5) | 3 (3)
HYPERTENSION (Vascular disorders) | 4 (4) | 1 (1) | 2 (2)
RETROPERITONEAL HAEMORRHAGE (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
AORTIC ATHEROSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ARTERIOVENOUS FISTULA THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
WOUND HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo.